CLINICAL TRIAL: NCT04145141
Title: A National Translational Science Network of Precision-based Immunotherapy for Primary Liver Cancer (PLC)
Brief Title: National Translational Science Network of Precision-based Immunotherapy for Primary Liver Cancer
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200006; 20-C-0006
Record Dates: First submitted 2019-10-29; First posted 2019-10-30 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01-16

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer; Cholangiocarcinoma
Keywords: Molecular Markers; Predictors for Response or Resistance to Immunotherapy; Sample Collection; Genetic Analysis; Natural History
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/ Cohort 1: Subjects with a diagnosis or suspicion of PLC

SUMMARY:
Background:

Primary Liver Cancer is the second most common cause of cancer-related death worldwide. It is the cancer with the fastest rising incidence and mortality in the United States. Researchers want to learn more about liver cancer to help them design better treatments.

Objective:

To better understand liver cancer.

Eligibility:

People ages 18 and older who have liver cancer and had or are planning to have immune therapy

Design:

Participants will be screened with a review of their medical records. They will be asked about their medical history and test results.

Participants will come to the NIH Clinical Center. During this visit, their medical records, test results, imaging studies, and tissue samples (if available) will be gathered. Participants will learn the results of a test to see if they have any mutations known to be connected to cancer. They will learn if there are treatment options for them. Participants will give blood, urine, and stool samples or rectal swabs.

Participants will not have follow-up visits just for this study. If they join another NIH research study and have visits for this other study, their medical records; test results; and blood, urine, and stool samples may be collected. This will occur about every 3 months. If they have a biopsy or surgery on another study or as part of treatment and there is leftover tissue, researchers would like to collect some of that tissue.

Participants will be contacted every 6 months by phone or e-mail. They will be asked about their health. They will provide any medical records, test results, and imaging studies.

Participants will be followed on this study for life.

DETAILED DESCRIPTION:
Background:

Primary liver cancer (PLC) is the 2nd most common cause of cancer-related death worldwide and the one cancer with the fastest rising incidence and mortality in the U.S. PLC consists of two main histological subtypes, i.e., hepatocellular carcinoma (HCC) and cholangiocarcinoma (CCA), in which diagnoses and treatment decisions are solely based on their baseline clinical features. However, whether these subtypes are truly distinct or share some fundamental features which can be pursued to improve clinical management is currently unclear. In addition, chronic liver diseases, due to complex etiologies such as viral hepatitis, alcohol consumption, chemicals, parasites or dietary factors, underlie and contribute to liver damage, increasing the risk of HCC and CCA development and progression. Consequently, PLC is clinically and biologically heterogeneous which has impeded biological assessment and clinical treatment.

Despite considerable efforts towards improving diagnosis and development of new treatment modalities, the improvement of PLC patient survival is minimal. For certain patients at early or intermediate disease stages, resection and percutaneous local ablation or Transarterial chemoembolization are available. However, the majority of patients present at advanced stages of disease, where the current gold standard of treatment is sorafenib, providing only a minimal improvement in survival time. PLC therefore remains among the most difficult-to-treat malignancies, with a 5-year survival rate of less than 15% in the United States. Thus, it is imperative that new treatment modalities are developed to limit cancer development and treat advanced PLC.

Immunotherapy (IO) is a promising new approach in PLC treatment. Alterations of the immune system, a component of the revised hallmarks of cancer, is recognized as a central player in carcinogenesis and cancer progression. Thus, strategies to inhibit or re-direct the immune response to the presence of tumors are currently being employed or developed. Immune-checkpoint inhibitors have shown promise in clinical trials of several solid tumors. Of particular note are monoclonal antibody-based therapy to block immune-inhibitory molecules, including programmed cell death protein-1 (PD-1), programmed cell death 1 ligand 1 (PDL-1) and cytotoxic T lymphocyte antigen 4 (CTLA4), which block anti-tumor T cell activity. However, the capacity of these therapies to reduce incidence and progression of PLC are still relatively unknown. Currently, several trials are underway to study the impact of immune checkpoint inhibitors as single agents or in combination with targeted therapy, on PLC development and outcome. Initial findings from Phase I/II clinical trials of PLC are promising but suggest that only certain patients respond to such treatment regimens while others do not or suffer from resistance/relapse. At the moment, it is difficult to determine which patient may benefit from immune therapy, due in large part to the lack of large comprehensive studies, biobank resources of specimens and biospecimen collection in clinical trial protocols, which deter our ability to understand and define critical genomic or genetic factors that contribute to patient response. Hence, we plan to collect PLC patient specimens and clinical data from those undergoing immunotherapies at NIH Clinical Center and a few extramural clinical sites to develop predictors for (a) response or resistance to immunotherapy and (b) acquired resistance to immunotherapy.

Objective:

To establish a biospecimen repository for genomic, genetic and epigenetic analysis to study the biology of PLC development and progression.

Eligibility:

Patients with histologically/ultrasound/imaging confirmed or suspicious lesions of HCC or CCA.

Patients with planned or a history of at least 1 dose of immunotherapy for HCC or CCA.

Age >= 18 years old at date of study consent

Design:

This will be a long-term multi-center study to comprehensively study patients with primary liver cancer (PLC).

Participants will provide clinical information (including medical history, clinical tests, imaging studies and reports, surgical pathology reports, genetic test results).

Tissue samples, blood, urine and fecal samples will be obtained from participants during this study.

Broad spectrum of scientific experiments, including genomics, metabolome, microbiome and immune monitoring will be performed.

Local physicians will be provided with test results of genomics panel evaluation (TruSight Oncology 500 (TSO-500).

Since long-term follow-up of individuals with PLC is a major feature of the study, local sites intend to maintain active contact with study subjects for as long as possible. Patients will be followed throughout the course of their illnesses, with particular attention to patterns of disease recurrence and progression, response to therapies and duration of responses. National death index data can also be utilized to obtain patient outcome information.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with histologically/ultrasound/imaging confirmed or suspicious lesions of HCC or CCA.
* Patients with planned or a history of at least 1 dose of immunotherapy for HCC or CCA.
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Age greater than or equal to 18 years old at date of study consent.

EXCLUSION CRITERIA:

- Patients with known HIV infection (as these patients may have abnormal test results which may confound the endpoints of this study)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To establish a biospecimen repository for genomic, genetic and epigenetic analysis to study the biology of PLC development and progression | 5 years
  Established biospecimen repository for genomic, genetic and epigenetic analysis to study the biology of PLC development and progression

SECONDARY OUTCOMES:
To estimate overall survival following immunotherapy for PLC | death
  Median amount of time subject survives from the beginning of immunotherapy.
To estimate 3 years progression-free survival following immunotherapy for PLC | 3 years
  Proportion of patients that have progressive disease after 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Tim F Greten, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (7):
- United States (7):
  - University of California, San Diego (UCSD), La Jolla, California
  - University of California, San Francisco (UCSF), San Francisco, California
  - Georgetown University, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.@@@@@@@@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.@@@@@@@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-C-0006.html